CLINICAL TRIAL: NCT06985446
Title: Assessment of Black Stains on Teeth in Relation to Salivary Parameters, Periodontal Health, and Body Mass Index in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozge Gungor, pHd, DDS, Assoc. Prof. Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AkdenizUıremkapıcı003
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Black Stains
Keywords: Salivary biomarkers; Child dental health; Body Mass Index (BMI); Oral health indices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black stain-positive (Experimental): The study group was named 'black stain-positive'
  Interventions: Other: Study Group:Black stain-positive
- Black stain-negative (Experimental): The control group was named 'black stain-negative'
  Interventions: Other: Control Group: Black stain-negative

INTERVENTIONS:
Other: Study Group:Black stain-positive — In children with black stains (BS+), we evaluated DMFT, dft, plaque index (Silness-Löe), gingival index (Löe-Silness), salivary pH, salivary flow rate, salivary buffering capacity, and body mass index (BMI).
  Arms: Black stain-positive
Other: Control Group: Black stain-negative — In healthy children without black stains (BS-), we assessed DMFT, dft, plaque index (Silness-Löe), gingival index (Löe-Silness), salivary pH, salivary flow rate, salivary buffering capacity, and body mass index (BMI).
  Arms: Black stain-negative

SUMMARY:
Objective The aim of this study is to compare salivary flow rate, salivary pH, salivary buffering capacity, plaque index, gingival index, DMFT/dft indices, and body mass index (BMI) in systemically healthy children aged 5-10 years with and without black stains (BS) in the oral cavity. By evaluating the differences between these two groups, we seek to better understand the effects of black stains on oral health and assess the relationship between BMI and these parameters. The findings may contribute to improved oral health management, preventive dentistry practices, and a deeper understanding of the association between obesity and oral health in children.

Methods This study will consist of two groups of systemically healthy children: those with black stains (BS group, n=50) and those without (non-BS group, n=50). Both groups will be examined to determine the d (decayed), f (filled), and t (missing) values for primary teeth (dft index) and D (decayed), M (missing), and F (filled) values for permanent teeth (DMFT index).

We will assess plaque index and gingival index using Silness-Löe (1963, 1967) criteria. Saliva samples will be collected under standardized conditions (at least 2 hours post-breakfast, between 9-11 AM, after rinsing with water) in an isolated dental unit with patients seated upright.

Salivary pH will be measured using pH strips (GC Saliva-Check BUFFER) from unstimulated saliva. We will categorize pH levels as: highly acidic (5.0-5.8, red), moderately acidic (6.0-6.6, yellow), or healthy (6.8-7.8, green).

For salivary flow rate measurement, stimulated saliva will be collected after paraffin chewing (5 minutes) and measured in mL/min.

Salivary buffering capacity will be evaluated using GC Saliva-Check BUFFER test pads and scored as: very low (0-5), low (6-9), or normal/high (10-12).

We will calculate Body Mass Index (BMI) as kg/m² and interpret results using age- and sex-specific percentiles.

Statistical analysis will compare all parameters between the two groups.

DETAILED DESCRIPTION:
This study will compare salivary parameters (pH, flow rate, buffering capacity), plaque index, gingival index, DMFT/dft indices, and BMI between healthy children aged 5-10 years with (n=50) and without (n=50) black stains (BS). Saliva samples will be collected under standardized conditions, oral health parameters will be recorded through clinical examinations, and statistical analysis will assess differences between the two groups. The aim is to evaluate the impact of BS on oral health and its potential association with BMI.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children (no chronic/acute systemic diseases)
* No antibiotic therapy within the last 3 months
* No use of medications affecting salivary flow (e.g., antihistamines, anticholinergics)
* No application of any plaque-disclosing agents recently
* Presence of clinically confirmed black stains on tooth surfaces
* No professional dental cleaning in the past 3 months
* No active caries lesions requiring immediate treatment

Exclusion Criteria:

* Presence of any systemic disease (e.g., diabetes, autoimmune disorders)
* Use of antibiotics or medications affecting salivary flow (e.g., antihistamines, antidepressants) in the last 3 months
* History of professional dental cleaning or scaling in the past 3 months
* Active dental caries requiring immediate treatment
* Diagnosed salivary gland disorders or xerostomia (chronic dry mouth)

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
DMFT index | 2 months
  To determine the DMFT index score, decayed teeth in permanent teeth are indicated as "D", lost teeth extracted due to decay are indicated as "M", and filled teeth are indicated as "F". The DMFT index is calculated by adding the D, M, F values and dividing them by the total number of permanent teeth. An increase in the calculated scores indicates that oral and dental health is negatively affected.
dft index | 2 months
  The dft Index is the calculated form of the DMFT index for primary teeth. When calculating the dft group index, missing teeth are not included in the calculation. Because it is difficult to diagnose the reason for the loss of primary teeth and there is a high probability of error. For this reason, the number of decayed and filled teeth is calculated during the examination. Decayed teeth are indicated with "d" and filled teeth with "f". The dft index is calculated by adding the d and f values and dividing them by the total number of permanent teeth. An increase in the calculated scores indicates that oral and dental health is negatively affected
Saliva pH | 2 months
  Salivary pH was measured using pH indicator strips. A low pH (<6.5) indicates an acidic environment and increases the risk of tooth demineralization and caries, whereas a high pH (>7.5) indicates an alkaline state, which may be linked to decreased bacterial activity but may also indicate systemic conditions.
Unstimulated salivary flow rate | 2 months
  Unstimulated salivary flow rate is measured by collecting unstimulated saliva over a period of time and calculating the volume per minute. A low flow rate (<0.1 mL/min) indicates hyposalivation, which increases the risk of caries and oral infection, while a high flow rate may be associated with conditions such as gastroesophageal reflux or medication effects.
Saliva buffering capacity | 2 months
  Saliva buffering capacity was measured using the GC Saliva Buffer Kit, which uses a scoring system based on color changes. A low buffering capacity indicates a higher risk of dental caries and enamel demineralization, whereas a high buffering capacity indicates better protection against acid attacks in the oral environment.
PIaque index (PI) | 2 months
  Based on Silness-Löe (1963, 1967) PI values, bacterial plaque and plaque thickness in direct contact with the marginal gingiva are evaluated. The evaluation is made with the Williams-marked University of Michigan 'O' periodontal probe, and PI values are recorded from a total of 4 surfaces of each tooth included in the study, namely mesial, distal, buccal and lingual. The averages of these values are calculated for each patient. The average scores obtained are evaluated in the 0-3 score range. An increase in the calculated scores indicates that periodontal health is negatively affected.
Gingival index (GI) | 2 months
  The degree of gingivitis is assessed using the Silness-Löe (1963, 1967) GI. The average of the measurements taken from four sides of the tooth determines the GI score of the tooth, and the average of the measurements of all teeth determines the individual's gingival index score. The scores obtained are evaluated in the range of 0-3. An increase in the calculated scores indicates that periodontal health is negatively affected.
Body Mass Index (BMI) | 2 months
  BMI is calculated by dividing weight (in kilograms) by the square of height (in meters) (kg/m²). In children, unlike adults, BMI is evaluated using age- and sex-specific percentile curves. An increase in BMI indicates a higher risk of obesity, which is associated with cardiovascular diseases, diabetes, and oral health problems such as periodontal disease and caries. A decrease in BMI may suggest undernutrition or growth retardation, potentially affecting immune function and dental development.
Percentile | 2 months
  Percentile is a statistical measure that indicates a child's BMI relative to other children of the same age and sex. It is determined using WHO (World Health Organization) or CDC growth charts.A high percentile (≥85th) indicates that the child is heavier than peers, increasing the risk of obesity and metabolic complications. A low percentile (<5th) suggests growth retardation or malnutrition risk, which may manifest as oral mucosal lesions or delayed tooth development.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Kapıcı, Research Assistant, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Faculty of Dentistry, Department of Pediatric Dentistry, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No